CLINICAL TRIAL: NCT01177280
Title: Prevalence of Potential Cytochrome P450 Pharmacokinetic Incident Drug-Drug Interactions Among Chronic Low Back Pain Patients Taking Opioid Analgesics and Associated Economic Outcomes
Status: Completed | Type: Observational
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Joseph Pergolizzi, MD, NEMA Research
Other Study IDs: CYP450cLBP4
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Low Back Pain
Keywords: retrospective chronic low back pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
This study explored the prevalence of DDEs in a chronic pain population with cLBP and associated healthcare utilization and costs using a healthcare claims database.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic low back pain patients
Sampling Method: Non-Probability Sample
Enrollment: 10000
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)